CLINICAL TRIAL: NCT05463120
Title: Minipuberty of Infancy and the Timing of Pubertal Development in Adolescence: a Follow-up of the Infant Feeding and Early Development (IFED) Cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000945; 000945-E
Record Dates: First submitted 2022-07-15; First posted 2022-07-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-18

CONDITIONS: Puberty
Keywords: Childhood; Growth; Adolescence; Hormone; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IFED-2: Children who participated in the IFED study as infants (2010-2014) and a parent/guardian will be enrolled in this follow-up study in childhood and followed for at least one year.

SUMMARY:
Background:

Earlier puberty is associated with adverse health throughout a person s life. The average age when puberty begins has been declining over the past decades in girls, and may also be declining in boys. The reasons for this shift are unknown.

Objective:

To determine whether internal (physical, hormonal) or external (feeding, environment) factors during infancy affect growth and the timing of puberty.

Eligibility:

Mothers (or other parent/guardian) and their children who completed the Infant Feeding and Early Development (IFED) study.

Design:

Participants will complete all activities at home for this natural history study.

Participant mothers will fill out two 15-minute questionnaires:

* One will be about themselves. They will answer questions about their body size in childhood, their puberty, and their pregnancies.
* The other will be about their child. They will answer questions about their child s puberty and lifestyle.

Child participants will fill out a questionnaire about their body changes during puberty. This will take 10 minutes.

Participants will be sent an electronic scale and a measuring tape. They will measure the child s weight, height, and waist and hip circumference. These numbers can be submitted online or by phone or mail.

Participants will receive a kit for collecting urine samples. Child participants will collect urine in a cup upon waking 4 days in a row. A special filter card is dipped in the cup then hung to dry. The dried cards will be mailed back.

Participants will allow researchers to access their child s medical records.

Questionnaires and body measurements will be repeated after 6 and 12 months. Urine sample collection will be repeated after 12 months.

All questionnaires can be done either online, by mail, or by phone on request.

DETAILED DESCRIPTION:
Study Description: Our overarching hypothesis is that endogenous and exogenous factors related to hypothalamic-pituitary-gonadal (HPG) axis activity during minipuberty of infancy are associated with childhood growth, the timing of pubertal development, and HPG axis activity in adolescence. To examine this hypothesis, we will conduct an observational follow-up study of children previously enrolled as infants in the Infant Feeding and Early Development (IFED) cohort. This follow-up study will be conducted remotely with data collection via email/online, mail and telephone by contractors at DLH, working on behalf of NIEHS.

Objectives: Primary Objective: To assess whether endogenous (e.g. hormone concentrations and size of hormone-sensitive organs) and exogenous (e.g. infant feeding method, exposure to endocrine disrupting chemicals) factors during minipuberty of infancy are related to a) growth, b) timing of pubertal development, and c) HPG axis activity in adolescence.

Endpoints: Primary Endpoints:

1. Height, weight and body mass index (BMI)
2. Onset of breast, pubic hair and/or genital development
3. Urinary metabolites of reproductive hormones (e.g. gonadotropins and sex steroids)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Completion of the original IFED study, defined as participants who did not withdraw from the study or were not withdrawn by the investigator prior to the end of original follow-up (up to 7 months in males and 9 months in females) and who provided at least the minimum number of blood samples (3 for boys, 4 for girls) across the original study period (N=283 eligible families).
2. Ability of subject and mother to understand and the willingness to review informed assent and consent documents, respectively, and indicate agreement to participate.

EXCLUSION CRITERIA:

We will not exclude any participants that meet the inclusion criteria from participating in the study overall or in any of the study procedures. We will collect information, via maternal report and linked medical records, on relevant medical diagnoses and the use of medications that may affect hormone levels, growth, and pubertal development. We may exclude participants with reported conditions or medication use (listed below) from analyses of some study aims or in sensitivity analyses.

Diagnoses/conditions:

* Central or peripheral precocious puberty
* Delayed puberty
* Growth hormone deficiency
* Stunted or delayed growth
* Idiopathic short stature
* Hypopituitarism
* Thyroid conditions, such as hyperthyroid, hypothyroid, Graves disease, Hashimoto's thyroiditis
* Genetic conditions, such as Prader-Willi syndrome, Turner syndrome, and Noonan syndrome

Medications:

* Gonadotropin-Releasing Hormone Agonists (e.g., leuprolide acetate (Lupron Depot), triptorelin (Triptodur), histrelin implant (Supprelin LA))
* Hormone therapy (e.g., testosterone, estrogen)
* Synthetic human growth hormone or IGF-1
* Synthetic thyroid hormone (e.g., levothyroxine)
* Anti-thyroid medications (e.g., methimazole, propylthiouracil) or radioactive iodine treatment

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The eligible population includes 283 children (136 girls, 147 boys), and their mothers or other parent/guardian, who completed the original IFED study, conducted when the children where 0-9 months of age (2010-2014).
Sampling Method: Non-Probability Sample
Enrollment: 566 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
To assess whether growth, timing of pubertal development, and hypothalamic-pituitary-gonadal (HPG) axis activity in childhood and adolescence are related to endogenous and exogenous endocrine-related factors during minipuberty of infancy. | Various time points in childhood/adolescence (study enrollment, 6-month and 12-month follow-up visits currently planned). We anticipate that children will be 8-12 years of age at enrollment (2022) and followed prospectively.
  1)Growth in height, weight and body mass index 2)Onset of pubic hair development, breast development (females), genital development (males) 3)Urinary concentrations of reproductive hormone metabolites (e.g., gonadotropins, estradiol, testosterone)

CONTACTS AND LOCATIONS:
Overall Officials: Dale P Sandler, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - National Institute of Environmental Health Sciences (NIEHS), Bethesda, Maryland
  - Social & Scientific Systems, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be shared with other researchers upon request. Plans for sharing data if requested are included in the study protocol.